CLINICAL TRIAL: NCT06868394
Title: Chronic Liver Disease and Radiation-induced Second Primary Liver Malignancy: a SEER Database Analysis 2010-2021
Brief Title: Chronic Liver Disease and Radiation-induced Second Primary Liver Malignancy
Status: Completed | Type: Observational
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, asmaa salama ibrahim, Resident physician of gastroenterology, Suez Canal University
Other Study IDs: H2730
Record Dates: First submitted 2025-02-26; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Chronic Liver Disease (CLD); Cancer; Liver Fibrosis
Keywords: chronic liver; SEER; Liver fibrosis; ISHAK score
MeSH Terms: conditions — Neoplasms; Liver Cirrhosis | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients with no to moderated liver fibrosis (ISHAK 0-4): They were subgrouped according to previous history of radiotherapy exposure into two groups. Both groups were followed up for 10 years to assess the risk of second primary malignancies. The investigators retrospectively analyzed the data.
  Interventions: Radiation: radiotherapy; Other: No intervention
- Patients with advanced or severe liver fibrosis (ISHAK 5-6): They were subgrouped according to previous history of radiotherapy exposure into two groups. Both groups were followed up for 10 years to assess the risk of second primary malignancies. The investigators retrospectively analyzed the data.
  Interventions: Radiation: radiotherapy; Other: No intervention

INTERVENTIONS:
Radiation: radiotherapy — The impact of previous radiotherapy exposure was studied on developing second primary malignancies.
Other: No intervention — This group received no radiotherapy

SUMMARY:
Cancer survivors are at a high risk to develop second primary malignancy (SPM) which constitutes a serious threat for them. Radiotherapy is the cornerstone for the management of many cancers as a locoregional treatment modality. Due to the low liver tolerance, cirrhotic patients are at a high risk of developing radiation-induced liver toxicities despite the modern safe radiation delivery techniques. Radiation damages cells through direct energy deposition and reactive free radical generation. Recent studies demonstrated a potential risk of SPMs following radiotherapy with further investigations for strategies to decrease radiation-induced SPMs. However, it is insufficiently addressed if developing liver SPMs is a serious adverse event following radiotherapy for cirrhotic patients. The aim of this study was to quantitatively assess the risk of gastrointestinal (GI) and liver SPMs following radiotherapy in patients with chronic liver disease.

DETAILED DESCRIPTION:
The SEER.stat software version 8.4.3 was used to obtain and analyze the data of patients with chronic liver disease diagnosed from 2010 to 2021. Using Ishak fibrosis score: F0-4 no to moderate fibrosis and F5-6 advanced or severe cirrhosis. patients were subgrouped according to the history of receiving radiotherapy for prior cancer treatment in two groups and excluded patients with unknown radiotherapy administration history. An MP-SIR session was used to calculate the Standardized Incidence Ratio (SIR) as Observed/Expected (O/E) with 95% confidence interval (CI). Significance was achieved at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients were classified according to fibrosis severity using the Ishak fibrosis score: F0-F4 (no to moderate fibrosis) and F5-F6 (advanced or severe cirrhosis) from 2010 to 2021.

Exclusion Criteria:

* Patients with unknown radiotherapy history or unknown fibrosis score or missing age data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Using the Surveillance, Epidemiology and End Results (SEER) database (17 Registries, 2000-2021, November 2023 Submission), maintained by the National Cancer Institute (NCI) containing a population-based cancer incidence and survival data from 17 registries covering approximately 28% of the U.S. population to extract the data of cancer patients with chronic liver disease diagnosed from 2010 to 2021. Patients were classified according to fibrosis severity using the Ishak fibrosis score: F0-F4 (no to moderate fibrosis) and F5-F6 (advanced or severe cirrhosis) from 2010 to 2021. Patients were stratified based on previous radiotherapy exposure into two groups; who received radiotherapy including beam radiation, radioactive implants, radioisotopes, combinations, or unspecified radiotherapy methods and patients who received no radiotherapy.
Sampling Method: Probability Sample
Enrollment: 20846 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The standardized incidence ratio and excess risk of developing gastrointestinal and liver second primary malignancies following radiotherapy exposure in patients with chronic liver disease (ISHAK 0-4) | from Jan, 2010 till Dec, 2021
  The surveillance, epidemiology and End Results (SEER) database was used to calculate the standardized incidence ratio (SIR) as Observed/Expected (O/E) and calculated the Excess absolute risk for multiple primary gastrointestinal and liver malignancies following radiotherapy exposure in patients with chronic liver disease (ISHAK 0-4)
The standardized incidence ratio and excess risk of developing gastrointestinal and liver second primary malignancies following radiotherapy exposure in patients with chronic liver disease (ISHAK 5-6) | from Jan, 2010 till Dec, 2021
  The surveillance, epidemiology and End Results (SEER) database was used to calculate the standardized incidence ratio (SIR) as Observed/Expected (O/E) and calculated the Excess absolute risk for multiple primary gastrointestinal and liver malignancies following radiotherapy exposure in patients with chronic liver disease (ISHAK 5-6)

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided